CLINICAL TRIAL: NCT02167685
Title: A Prospective Observational Study for the Long-term Follow-up of Subjects Previously Enrolled in Selected Clinical Studies of CMX001.
Brief Title: The Chimerix CMX001 Registry
Acronym: CMX001
Status: Terminated | Type: Observational
Why Stopped: terminated due to low enrollment rate
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CMX001-333
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Outcomes; Survival Rates
MeSH Terms: interventions — brincidofovir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CMX001: Subjects who have previously participated in CMX001-301 or other CMX001 study.
  Interventions: Drug: CMX001

INTERVENTIONS:
Drug: CMX001
  Other Names: Brincidofovir

SUMMARY:
The prospective observational study is to establish a registry database to evaluate the potential impact of prior treatment with CMX001 on the long-term incidence of specific events, such as outcomes, late CMV and other Double-stranded DNA virus associated events, s well as survival rates in subjects previously enrolled in selected clinical studies of CMX001. Each Registry participant will be followed for a period of approximately 3 years from their enrollment in the Registry.

ELIGIBILITY:
Inclusion Criteria:

* Have previously completed study CMX001-301 through the Week 24 visit, or participated in another qualifying clinical study with CMX001.
* Willing and able to understand and provide written informed consent to participate in this observational study
* Willing and able to participate in all required study activities for the entire duration of the observational study (i.e., agreeable to being contacted at periodic intervals over the course of approximately 10 years following the completion of study CMX001-301 or other qualifying clinical study.

Exclusion Criteria:

* None

Ages: 6 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects previously enrolled in selected clinical studies of CMX001
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Time to all-cause mortality | 10 years
  evaluate the potential impact of prior treatment with CMX001 on the long-term incidence of specific events, such as the development of new malignancies and late cytomegalovirus (CMV)-associated events, as well as survival rates in subjects previously enrolled in selected clinical studies of CMX001

CONTACTS AND LOCATIONS:
Locations (51):
- United States (47):
  - University of California San Diego, La Jolla, California
  - St. Vincent Medical Center, Los Angeles, California
  - Children's Hospital of LA, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Childrens Hospital of Colorado, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - University of Colorado Hospital/Health Science Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital/Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children Mercy Hospital and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Hackensack, Hackensack, New Jersey
  - Mt Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weil Cornell Medical Center, New York, New York
  - Albert Einstein Cancer Center at Montefiore Medical Park, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University Baptist Center, Winston-Salem, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Allegheny-Singer Cancer Institute, Pittsburgh, Pennsylvania
  - St. Judes Children's Hospital, Memphis, Tennessee
  - Baylor Cancer Center, Dallas, Texas
  - University of Texas-MD Anderson, Houston, Texas
  - Methodist Healthcare System, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - Intermountain Center for Hematological Malignancies, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Centre Hospitalier Unversitaire Sart, Liège
- Canada (2):
  - University of Toronto, Toronto, Ontario
  - Hopital Maisonneuve-Rosement, Montreal, Quebec